CLINICAL TRIAL: NCT05968742
Title: Mechanisms Underlying the Variation in Rate and Levels of Gingival Inflammatory Responses Among the Human Population
Brief Title: Variation in Gingival Inflammatory Responses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Jeffrey McLean, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00016247; R01DE031470 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Gingivitis
Keywords: Experimental Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective clinical study using the experimental gingivitis model. Split Mouth design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Study participants abstain from oral hygiene on a select set of four teeth for a period of 21 days.
  The use of a custom made acrylic intraoral stent (mouthguard) will be used to protect teeth on designated test sides for each study participant during normal oral hygiene (approximately 4 minutes each day: 2 times for 2 minutes) throughout the induction phase (Day 0-21).
  Interventions: Behavioral: Abstinence of oral hygiene on select teeth

INTERVENTIONS:
Behavioral: Abstinence of oral hygiene on select teeth — Study participants abstain from oral hygiene on a select set of four teeth for a period of 21 days
  Other Names: Split Mouth Experimental Gingivitis

SUMMARY:
The aim of this NIH National Institute of Dental and Craniofacial Research (NIDCR) funded study is to identify molecular mechanisms underlying observed variations in human responses to natural accumulation and maturation of dental plaque.

DETAILED DESCRIPTION:
This study will employ the split-mouth Experimental Gingivitis model where healthy study participants are asked to abstain from oral hygiene on a select set of teeth (test teeth) for a period of 21 days. The study consists of 3 phases; Hygiene Phase (Day -14-0), Experimental Induction Phase (Day 0-21), and Resolution Phase (Day 21-35). Abstaining from oral hygiene on the test teeth will result in the natural accumulation and maturation of dental plaque (a bacterial biofilm) on the tooth surface which will in induce a host inflammatory response. By investigating the onset of microbially induced inflammation directly in humans using this highly utilized and well-described experimental gingivitis model, the research community are able to better understand the host-microbial interactions during the initiation, induction of host response, and resolution of mucosal inflammation at the molecular level. The investigators central hypothesis is based on our previous experimental gingivitis studies conducted here at the University of Washington Bamashmous et al. Human Variation in Gingival Inflammation PNAS 2021 and NCT03750955. The investigators hypothesize that specific clinical inflammatory response phenotypes (High, Low and Slow responders) are dependent upon both microbial factors regulating the subgingival plaque growth and maturation rate as well as host factors regulating the human gingival inflammatory mediator levels and type.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 18-35 years
* Good general health, ASA I (healthy with no systemic conditions)
* No clinical signs of gingival inflammation at > 90% of sites observed (whole mouth) (< 10% of sites with GI of < 2 and no sites with a score of 3; < 10% sites with BOP +).
* Probing depth (PD) ≤ 3.0 mm (Whole Mouth)
* Attachment loss (AL) = 0 mm (Whole Mouth)
* Gingival health at Visit 2 (Day 0) for study sites (Test/Control teeth): Average Gingival Index (GI) ≤ 0.1 with no site having a score of 3 and bleeding on probing (BOP)(-)
* Never smokers
* The ability to understand and communicate with the examiner.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Medical condition which requires premedication prior to dental treatments/visits
* Subjects unable or unwilling to sign the informed consent form
* History of periodontal disease
* History of systemic inflammatory or immune conditions, Diabetes
* Use of antibiotic or anti-inflammatory drugs within 30 days of enrollment
* Self-reported pregnancy, planned pregnancy during the planned study commitment, and/or breastfeeding at the time of screening.
* Concurrent orthodontic treatment
* Untreated carious lesions and/or inadequate restorations on maxillary posterior teeth
* Participation in any other clinical study or test panel within 1 week prior to enrollment into this study
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates
* Orthodontic bands, appliances, or crowns and bridges, or removable partial dentures affecting the maxillary posterior teeth
* Missing tooth/teeth within the study sites test and control
* History of allergy to common dentifrice ingredients
* Immune-compromised individuals (for example: HIV, AIDS, and immune-suppressive drug therapy)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of clinical responder types | Day 0 to Day 21
  Identification of clinical responder types through comparative analysis of the levels of clinical parameter for Bleeding on Probing Index (% BOP) at Day 14 of the plaque overgrowth/induction phase measured by calibrated examiners.

SECONDARY OUTCOMES:
Change in relative abundance of bacteria | Day 0 to Day 21
  The rate of change in relative abundance of gram positive Firmicutes bacteria compared to that of gram negative Bacteroidetes bacteria through the plaque overgrowth/induction phase (Day 0-21) assessed through 16S rRNA and Metagenomic Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S McLean, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bamashmous S, Kotsakis GA, Kerns KA, Leroux BG, Zenobia C, Chen D, Trivedi HM, McLean JS, Darveau RP. Human variation in gingival inflammation. Proc Natl Acad Sci U S A. 2021 Jul 6;118(27):e2012578118. doi: 10.1073/pnas.2012578118. PMID 34193520